CLINICAL TRIAL: NCT07041281
Title: Spironolactone to Improve Pregnancy-Associated Hypertension Trajectories
Acronym: IMPACT-HT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Michael C. Honigberg, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P001195; 25SFRNPCKMS1463898 (Other Grant/Funding Number: American Heart Association); STUDY25060149 (Other: University of Pittsburgh Institutional Review Board)
Record Dates: First submitted 2025-06-11; First posted 2025-06-27 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Preeclampsia; Gestational Hypertension
Keywords: preeclampsia; gestational hypertension; spironolactone; blood pressure; hypertension; pregnancy; echocardiography
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Hypertension | interventions — Spironolactone

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, placebo-controlled trial of low-dose spironolactone versus placebo in women with pre-pregnancy overweight/obesity who develop de novo hypertensive disorders of pregnancy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo: Control (Placebo Comparator): Participants with Hypertensive disorders of pregnancy will receive placebo equivalent capsules to self-administer daily over the 12-week duration of the study treatment.
  Interventions: Drug: Placebo tablet to match spironolactone
- Treatment: Spironolactone (Experimental): Participants with hypertensive disorders of pregnancy will receive 25mg capsules of spironolactone to self-administer daily over the 12-week duration of the study treatment.
  Interventions: Drug: spironolactone 25 mg orally once daily

INTERVENTIONS:
Drug: spironolactone 25 mg orally once daily — Participants with hypertensive disorders of pregnancy will receive 25mg capsules of spironolactone to self-administer daily over the 12-week duration of the study treatment.
  Arms: Treatment: Spironolactone
Drug: Placebo tablet to match spironolactone — Participants with Hypertensive disorders of pregnancy will receive placebo equivalent capsules to self-administer daily over the 12-week duration of the study treatment.
  Arms: Placebo: Control

SUMMARY:
The hypertensive disorders of pregnancy (preeclampsia and gestational hypertension) are associated with increased long-term maternal risk of developing cardiovascular disease. Recent evidence suggests that activation of the mineralocorticoid receptor promotes ongoing susceptibility to hypertension in women following hypertensive disorders of pregnancy. In addition, women with overweight/obesity are at increased risk for progression to chronic hypertension after experiencing hypertensive disorders of pregnancy. Among women with hypertensive disorders of pregnancy and pre-pregnancy overweight/obesity, the investigators will conduct a randomized trial to test the effect of pharmacologically blocking the mineralocorticoid receptor for three months after delivery on blood pressure and cardiac remodeling at nine months postpartum.

DETAILED DESCRIPTION:
The hypertensive disorders of pregnancy (HDP, e.g., gestational hypertension and preeclampsia) are a leading cause of maternal and infant morbidity and mortality and are associated with increased long-term risk of maternal atherosclerotic cardiovascular disease (CVD) and heart failure. The American College of Cardiology and American Heart Association now recognize the HDP as a sex-specific CVD risk factor to guide prescription of preventive statin therapy. Beyond this focused recommendation, however, targeted strategies for CVD risk reduction in women with HDP are not yet established. Maternal overweight/obesity is a risk factor for accelerated progression from HDP to chronic hypertension, a key mediator of heightened long-term CVD risk in women with a history of HDP, and for adverse cardiac remodeling in pregnancy. Recent preclinical evidence suggests that the HDP induce heightened vascular smooth muscle cell mineralocorticoid receptor (MR) sensitivity that persists postpartum, promoting chronic hypertension and CVD. In addition, the recent POP-HT trial suggested that blood pressure control in the very early postpartum period has long-lasting effects on the risk of chronic hypertension and cardiac remodeling in women after HDP. Integrating these lines of evidence, the investigators hypothesize that short-term pharmacologic blockade of the MR in the early postpartum period after HDP will yield long-term maternal cardiovascular benefits in women with overweight/obesity. To test this hypothesis, the investigators will compare a strategy of adding low-dose spironolactone, a breastfeeding-compatible MR antagonist, or placebo to usual care for 3 months following delivery with HDP. This multi-site trial will randomize 204 women with HDP and pre-pregnancy overweight/obesity delivering at Massachusetts General Hospital, Brigham and Women's Hospital, and the University of Pittsburgh-Magee Womens Hospital. The investigators will test the effect of short-term adjunctive postpartum spironolactone on 24-hour ambulatory blood pressure (Aim 1) and postpartum cardiac remodeling by echocardiography (Aim 2) at 9 months postpartum (i.e., 6 months after completion of study treatment).

ELIGIBILITY:
Inclusion Criteria:

* Females aged ≥18 years
* Antepartum-onset HDP (gestational hypertension or preeclampsia) without pre-pregnancy chronic hypertension
* BMI ≥25 kg/m2 prior to pregnancy or in the first trimester
* Requirement for antihypertensive medication on postpartum discharge
* Ability to provide informed consent

Exclusion Criteria:

* LV ejection fraction <50% or history of clinical heart failure with reduced or preserved ejection fraction
* Hypertrophic or other genetic cardiomyopathy
* Hyperkalemia: potassium >5.3 mEq/L
* BMI at screening ≥50 kg/m2 (to ensure accurate BP measurement and adequate echocardiographic images for analysis)
* Pre-pregnancy diabetes
* Estimated glomerular filtration rate (eGFR) <60mL/min/1.73 m2
* Cirrhosis
* Primary aldosteronism
* Intention to become pregnant within 9 months
* Active substance abuse
* Other serious medical illnesses or concerns about protocol adherence/ mortality within 9 months
* Participation in another interventional clinical study
* Hypersensitivity to spironolactone
* Addison's disease
* Concomitant use of eplerenone or finerenone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-12-02 (Estimated); Study Completion 2029-03-02 (Estimated)

PRIMARY OUTCOMES:
Mean 24-hour ambulatory diastolic blood pressure | 36 weeks
  24-hour BP monitoring will be performed as part of end-of-study assessments using a validated ambulatory BP monitor.

SECONDARY OUTCOMES:
Left ventricular relative wall thickness (main echocardiographic outcome) | Baseline and 36 weeks
  Relative wall thickness is calculated as 2*posterior wall thickness/LV end-diastolic diameter as measured by transthoracic echocardiography.
Mean 24-hour ambulatory systolic blood pressure | 36 weeks
  24-hour BP monitoring will be performed as part of end-of-study assessment using a validated ambulatory BP monitor. Mean 24-hour systolic BP will be calculated from the device data.
Mean diurnal ambulatory systolic blood pressure | 36 weeks
  24-hour BP monitoring will be performed as part of the end-of-study assessment using a validated ambulatory BP monitor. Mean diurnal systolic BP will be calculated from the device data.
Mean diurnal ambulatory diastolic blood pressure | 36 weeks
  24-hour BP monitoring will be performed as part of the end-of-study assessment using a validated ambulatory BP monitor. Mean diurnal ambulatory diastolic blood pressure will be calculated from the device data
Mean nocturnal ambulatory systolic blood pressure | 36 weeks
  24-hour BP monitoring will be performed as part of the end-of-study assessment using a validated ambulatory BP monitor. Mean nocturnal ambulatory systolic blood pressure will be calculated from the device data.
Mean nocturnal ambulatory diastolic blood pressure | 36 weeks
  24-hour BP monitoring will be performed as part of the post-treatment assessments using a validated ambulatory BP monitor. Mean nocturnal ambulatory diastolic blood pressure will be calculated from the device data.
Measured systolic blood pressure | Baseline, 2 weeks, 12 weeks, and 36 weeks
  At each visit, BP will be measured by study staff three times at one-minute intervals in accordance with multi-society guidelines for accurate measurement of blood pressure. The first measurement will be discarded, and the average of the second and third measurements will be recorded as the measured BP at each study visit.
Measured diastolic blood pressure | Baseline, 2 weeks, 12 weeks, and 36 weeks
  At each visit, BP will be measured by study staff three times at one-minute intervals in accordance with multi-society guidelines for accurate measurement of blood pressure. The first measurement will be discarded, and the average of the second and third measurements will be recorded as the measured BP at each study visit.
Readmission for hypertension | Through study completion (36 weeks post-randomization)
  Postpartum readmission for hypertension will be captured.
All-cause readmission | Through study completion (36 weeks post-randomization)
  All postpartum readmission will be captured
Daily defined doses of antihypertensive medication | Baseline, 2 weeks, 12 weeks, and 36 weeks
  Daily defined doses of antihypertensive medication will be quantified in accordance with the World Health Organization classification.
Time to discontinuation of all non-study drug antihypertensive medications | Through study completion (36 weeks post-randomization)
  All medication changes made by treating clinicians will be captured.
Escalation of antihypertensive regimen | Through study completion (36 weeks post-randomization)
  All medication changes made by treating clinicians will be captured.
Ratio of mitral E velocity to e' [E/e'] | Baseline and 36 weeks
  E/e', a measure of diastolic function, will be measured by transthoracic echocardiography.
Early diastolic septal mitral annular velocity [septal e'] | Baseline and 36 weeks
  Septal e', a measure of diastolic function, will be measured by transthoracic echocardiography using tissue Doppler
Peak tricuspid regurgitant jet velocity | Baseline and 36 weeks
  Peak tricuspid regurgitant jet velocity, a measure of diastolic function, will be measured by transthoracic echocardiography using continuous wave Doppler
Left atrial volume index | Baseline and 36 weeks
  Left atrial volume index will be measured by transthoracic echocardiogarphy using the biplane method and indexed for body surface area.
Ratio of E to A [E/A] | Baseline and 36 weeks
  E/A, a measure of diastolic function, will be measured by transthoracic echocardiography.
Left ventricular mass index | Baseline and 36 weeks
  Left ventricular mass will be calculated from transthoracic echocardiogarphy using the Devereux formula and indexed for body surface area
Left ventricular ejection fraction | Baseline and 36 weeks
  Left ventricular ejection fraction will be measured by transthoracic echocardiogarphy using the biplane method.
Left atrial reservoir strain | Baseline and 36 weeks
  Left atrial strain, a sensitive measure of end- diastolic pressure and atrial remodeling, will be quantified using TOMTEC.
Peak global longitudinal strain | Baseline and 36 weeks
  Left ventricular global longitudinal strain, a measure of subclinical cardiac dysfunction, will be quantified using TOMTEC.
Interventricular septal wall thickness | Baseline and 36 weeks
  Interventricular septal wall thickness will be measured by transthoracic echocardiography from the parasternal long axis view.
Posterior wall thickness | Baseline and 36 weeks
  Posterior wall thickness will be measured by transthoracic echocardiography from the parasternal long axis view.
High-sensitivity cardiac troponin I | Baseline, 12 weeks, and 36 weeks
  High-sensitivity cardiac troponin will be measured using standard clinical assays.
N-terminal pro-B-type natriuretic peptide | Baseline, 12 weeks, and 36 weeks
  NT-proBNP will be measured using standard clinical assays.
Urine microalbumin/creatinine | 2 weeks, 12 weeks, and 36 weeks
  Urine microalbumin/creatinine will be measured using standard clinical assays.
Activin A | Baseline, 2 weeks, 12 weeks, and 36 weeks
  Activin A will be measured by ELISA.
Soluble fms-like tyrosine kinase receptor-1 | Baseline, 2 weeks, 12 weeks, and 36 weeks
  sFlt-1 will be measured by ELISA.
Placental growth factor | Baseline, 2 weeks, 12 weeks, and 36 weeks
  Placental growth factor will be measured by ELISA.
Procollagen type I carboxyterminal propeptide | Baseline, 12 weeks, and 36 weeks
  PICP will be measured by enzyme immunoassay.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Pittsburgh Magee-Womens Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No